CLINICAL TRIAL: NCT06808945
Title: Preoperative PREhabilitation in Patients Planned for LIVER Transplantation (PRELIVERT)
Brief Title: Preoperative Prehabilitation in Patients Planned for Liver Transplantation
Acronym: PRELIVERT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Rijndam Revalidatiecentrum (Unknown); Capri Hartrevalidatie (Unknown)
Responsible Party: Principal Investigator, Roeland F. de Wilde, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL85306.078.23
Record Dates: First submitted 2024-11-25; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Liver Transplant; Complications; Physical Inactivity
Keywords: prehabilitation; liver transplant
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Home based prehabilitation (Experimental): Participants will be subjected to a training period of eight weeks of a home-based multimodal prehabilitation program. The program consists of an exercise program, nutritional support, smoking cessation and psychological counselling.
  Interventions: Other: Prehabilitation program

INTERVENTIONS:
Other: Prehabilitation program — Participants will be subjected to an eight week home-based multimodal prehabilitaiton program. The program consists of an exercise program, nutritional support, smoking cessation and psychological counselling.

SUMMARY:
The objective of this study is to determine the feasibility and effectiveness of a home-based multimodal prehabilitation program in patients anticipated to be waitlisted for LT. Patients will participate in an eight week prehabilitation program consisting of physical exercise, nutritional support, smoking cessation and psychological counselling.

DETAILED DESCRIPTION:
Rationale: Patients who qualify for liver transplantation (LT) are mostly frail due to their underlying liver disease. Frailty is comprised by a decreased functional capacity, impaired aerobic capacity, and sarcopenia. It is well known that frailty leads to both increased pre- and post-transplantation morbidity as well as mortality. For various surgical populations prehabilitation was demonstrated to be feasible, effective, and to improve surgical outcomes. Few studies on this subject have been conducted in the patient population awaiting liver transplantation.

Objective: The primary objective is to determine the feasibility of a semi-supervised homebased prehabilitation program for patients to be waitlisted for LT. The secondary objectives are to assess the effectiveness of this program and possible improvements of surgical outcomes (e.g. less complications, faster recovery, and shorter length of hospital stay).

Study design: This is a multi-centre, single arm, prospective cohort (pilot) study. It will take place at the Erasmus Medical Center in Rotterdam, the Netherlands.

Study population: Adult patients who are anticipated to be waitlisted for LT, who have no contra-indications to physical exercise training.

Intervention: Patients will participate in an eight-week semi-supervised home based prehabilitation program. This program consists of physical exercise, nutritional support provided by a dietician, smoking cessation, and psychological counselling. The program will be personalized and consists of two training sessions per week. Through the Oefenportaal platform the physical therapist will supervise the exercises and monitor patients' adherence to the program.

Main study parameters/endpoints: The main study parameter/endpoint is the feasibility of the prehabilitation program (program satisfaction, compliance, and percentage of patients willing to participate in the prehabilitation program). A secondary outcome is the effectiveness of the program. Furthermore, postoperative outcomes after 30 days will be collected.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients will participate in an eight-week prehabilitation program prior to anticipated LT. The prehabilitation sessions take approximately 3-5 hours per week. To lower the burden for patients, the majority of the program takes place at home using digital tools. During the first week patients are seen at the Erasmus MC for an intake (about 60 minutes). All study appointments will be combined with regular appointments for screening if possible. Furthermore, patients are expected on-site at the start and after completion of the prehabilitation program to undergo measurements (90 minutes). Also, they have to complete questionnaires at home three times total (two times 20 minutes, one time 10 minutes).

Since the prehabilitation program is based on existing care, we expect minimal risks for the patients. Participants are anticipated to benefit from the pilot prehabilitation program considering a better physical fitness and a behavioural change towards a healthier lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years,
* Anticipated waitlisting for LT,
* Speaks the Dutch language,
* Understands the purpose of the study and has given written informed consent.

Exclusion Criteria:

* Experienced a major adverse cardiovascular event in the past six months,
* Experienced a cerebrovascular incident in the past six months,
* Medical history of an uncontrolled heart rhythm disorder,
* Hepatic encephalopathy grade 3 or 4,
* Acute liver failure,
* Acute-on-chronic liver failure,
* Hospitalization at start of the study.
* Non-treated esophageal varices (i.e., no previous variceal eradication endoscopy or adequately dosed NSBB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Program satisfaction | At completion of the prehabilitation program (8 weeks after baseline/screening for LT)
  Self-designed questionnaire score (score between 1-10, higher score means higher satisfaction)
Program compliance | At completion of the prehabilitation program (8 weeks after baseline/screening for LT)
  Number of sessions that patient participates in the fitness training, the counselling on nutrition, smoking cessation and psychosocial sessions will be registered.
Percentage of patients willing to participate in the prehabilitation program | At the outpatient clinic, when patients make their appointment for screening for LT
  It will be registered which patients are willing and not willing to participate

SECONDARY OUTCOMES:
Aerobic capacity | At start of the program, when patients are admitted for screening, they will perform a CPET as baseline. After eight weeks of home-based training the CPET will be reassessed.
  A cardiopulmonary exercise test (CPET) will be performed by participants to determine their aerobic capacity pre-intervention and at the end of the program. The following outcomes will be assessed: VO2 at the VAT (ml/kg/min)
Sarcopenia | At baseline (before start prehabilitation program) and after eight weeks.
  Body composition will be determined by bioelectrical impedance analysis at baseline and after eight weeks. Also patients will be asked to fill out a sarcopenia specific questionnaire: the SARC-F.
Anthropometry | At baseline (before start prehabilitation program) and after eight weeks.
  Body mass and body height will be measured with a calibrated electronic scale and e metric measuring tape with a wall stop.
Functional capacity | At baseline (before start prehabilitation program) and after eight weeks.
  Patients are asked to walk as many meters as possible in a time period of 6 minutes.
Functional mobility | At baseline (before start prehabilitation program) and after eight weeks.
  Functional mobility will be assessed using the 30-second chair stand test.
Physical activity level | At baseline (before start prehabilitation program) and after eight weeks patients will wear the ActiGraph accelerometer for 7 days.
  ActiGraph GTx3+ accelerometer: average time per day (min) spend in moderate-to-vigorous activity, light physical activity and sedentary behaviour Futhermore patients will be asked to monitor the amount of steps taken per day using the 'Oefenportaal platform'
Hand grip strength | At baseline (before start prehabilitation program) and after eight weeks.
  Hand dynamometer (kg)
Quadriceps strength | At baseline (before start prehabilitation program) and after eight weeks
  Biodex dynamometer (Peak torque to body weight extension + Work fatigue)
Quality of life assessment | At baseline (before start prehabilitation program) and after eight weeks
  Questionnaire
Perceived fatigue assessment | At baseline (before start prehabilitation program) and after eight weeks
  Questionnaire
Postoperative outcomes up to 30 days post LT assessment | Through study completion (30 days after LT)
  All surgical relevant postoperative outcomes up to 12 months post LT are recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No